CLINICAL TRIAL: NCT05684640
Title: A Single and Multiple Dose Study of Rodatristat Ethyl in Healthy Subjects to Evaluate the Effect of Food, and the Safety, Tolerability, and Pharmacokinetics of a Supratherapeutic Dose of Rodatristat Ethyl
Brief Title: A Single and Multiple Dose of Rodatristat Ethyl in Healthy Adult Subjects to Evaluate the Effect of Food and Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altavant Sciences GmbH (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RVT-1201-1006
Record Dates: First submitted 2022-11-07; First posted 2023-01-13 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Healthy
MeSH Terms: interventions — rodatristat

STUDY DESIGN:
Intervention Model Description: Single and multiple dose
Who Masked: Participant, Investigator
Masking Description: There are 2 parts to the study. Part one is an open label parallel study and Part 2 is a randomized double-blind placebo controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rodatristat ethyl (Experimental): Part One: is 600 QD
  Interventions: Drug: Rodatristat Ethyl
- Placebo (Placebo Comparator): Part Two: Placebo match for Rodatristat ethyl
  Interventions: Drug: Rodatristat Ethyl; Drug: Placebo

INTERVENTIONS:
Drug: Rodatristat Ethyl — Tablets, Oral, 600mg, QD
Drug: Placebo — Tablets, Oral, 0mg, BID
  Arms: Placebo

SUMMARY:
This is a single and multiple dose food effect study of rodatristat ethyl in healthy subjects

DETAILED DESCRIPTION:
This is a two-part Phase 1 study. Part 1 is a single dose, randomized, open label, parallel, single site study designed to evaluate the effect of a high fat meal on the PK of rodatristat ethyl, rodatristat and metabolite(s). Part 2 is a randomized double-blind, placebo-controlled study to evaluate the safety and tolerability of repeat supratherapeutic dose of rodatristat ethyl when administered twice daily with a standard meal.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females aged 18 to 55 years, inclusive.
2. A male subject is eligible to participate if he does not have a female partner who is pregnant or who intends to become pregnant during the study. Male subjects must agree to use contraception starting at Screening, during the treatment period, and for at least 100 days after the last dose of study drug, and refrain from donating sperm during this period.
3. Female subjects of childbearing potential must agree to use contraception starting at Screening, during the treatment period, and for at least 4 weeks after the last dose of study drug.
4. Body mass index (BMI) ≥ 18 kg/m2 and ≤ 30 kg/m2.
5. Willing and able to give written informed consent and to comply with the requirements of the study for its duration.

Exclusion Criteria:

1. As determined by the Investigator, any known pre existing medical or psychiatric condition that could interfere with the subject's ability to provide informed consent or participate in study conduct, or that may confound study findings including, but not limited to a history of clinically significant gastrointestinal, hematologic, renal, hepatic, bronchopulmonary, neurological, psychiatric, or cardiovascular disease, including

   1. History of Gilbert's Syndrome
   2. History of depression
   3. History of any allergy that, in the opinion of the Investigator, contraindicates participation in the trial
2. Positive pregnancy test at Screening or Check-in.
3. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at Screening) of 50 mL to 499 mL of blood within 30 days or more than 499 mL within 56 days prior to starting study drug.
4. Participation in an investigational drug, vaccine, or device study within 30 days before study drug administration or 90 days for a biologic study.
5. Clinically significant ECG abnormalities.
6. Abnormal blood pressure, either low (defined as < 90 mmHg systolic and/or < 50 mmHg diastolic) or high (defined as > 140 mmHg systolic and/or > 90 mmHg diastolic) at Screening or prior to starting study drug.
7. Clinically significant abnormalities in laboratory test results, as determined by the Investigator, (including hepatic and renal panels, complete blood count, coagulation, chemistry panel, and urinalysis) at Screening or Check-in.

   1. Positive serology for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
   2. Estimated glomerular filtration rate < 90 mL/min/1.73 m2 at Screening, calculated using the Modification of Diet in Renal Disease (MDRD) formula.
   3. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) values greater than upper limit of normal (ULN).
   4. Positive urine test for drugs of abuse at Screening or Check-in.
   5. Positive alcohol test (breath, saliva, or urine) at Screening or Check-in.
   6. Positive pregnancy test at Screening or Check-in.
8. Use of prescription or nonprescription drugs, (with exception of contraceptive and acetaminophen allowance), including high dose vitamins, dietary supplements (including St. John's Wort) within 14 days or 5 half lives of the prescription or nonprescription drug (whichever was longer) prior to the first dose of study drug, through to the final follow-up visit.
9. Consumption of grapefruit or Seville oranges or their juices within the 7 days prior to dosing until collection of the final PK sample.
10. Use of medications associated with QT prolongation within 30 days prior to dosing and during the study.
11. Subjects unable to abstain from alcohol for 72 hours prior to the start of dosing through collection of the final PK sample.
12. Subjects with a clinical history of or current alcohol abuse defined as an average weekly intake of more than 21 units for males or 15 units for females (1 unit = 340 mL beer, 115 mL wine, or 43 mL spirits).
13. Subjects with a clinical history of or current illicit drug use which, in the opinion of the Investigator, would interfere with the subject's ability to complete the study.
14. Subjects unable to abstain from caffeine, xanthine, or strenuous exercise for 72 hours prior to dosing.
15. Subjects who have smoked or used tobacco- or nicotine containing products within 3 months prior to the Screening visit and who are unwilling to refrain from smoking, tobacco use, or use of nicotine products for the entire duration of the study.
16. Employed as site personnel directly involved with this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Part 1 will evaluate the effect of a high-fat meal on the PK of rodatristat ethyl, rodatristat, and its metabolite(s) following single-dose administration of a rodatristat ethyl 600 mg dose | 6 Days
  Measure Rodatristat, rodatristat ethyl, and its metabolite(s): Maximum plasma concentration Cmax, area under the plasma concentration-time curve from time zero (predose) to the last detectable time point.
Part 2 will assess the PK of rodatristat ethyl, rodatristat, and metabolite(s) following multiple repeat doses of rodatristat ethyl at a supratherapeutic level | 11 Days
  Measure PK parameters, area under the concentration time curve over the dosing interval.

SECONDARY OUTCOMES:
Part 1 will also evaluate the effect of a high-fat meal on other PK parameters of rodatristat ethyl, rodatristat, and its metabolites | 6 Day
  Measure PK parameters: time to maximum concentration (tmax).
Part 1 will also evaluate the effect of a high-fat meal on other PK parameters of rodatristat ethyl, rodatristat, and its metabolites | 6 Day
  Measure elimination of half life (t 1/2)
Part 2 will also assess the effect of a supratherapeutic dose of rodatristat ethyl on plasma 5 hydroxyindoleacetic acid (5 HIAA) concentrations | 11 Days
  Measure changes from baseline in plasma 5-HIAA concentrations from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hunt, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Development, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No